CLINICAL TRIAL: NCT05573152
Title: Pre Warming Protocol Implementation Strategy in the Operation Room Routine
Brief Title: Pre Warming Protocol Implementation in Operation Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Parecer 699.971
Record Dates: First submitted 2015-06-17; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Hypothermia
Keywords: Body Temperature; Hypothermia
MeSH Terms: conditions — Hypothermia | interventions — Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nursing (Experimental): Nursing Group (Nurse): the nursing team will use of the warming device air flow device from the moment the patients enter the operating room until anesthesia induction. The warming device will be set up connected to the patient and to the motor with the activation of the system at 43°C by the nursing team. The monitoring of the times since the entrance of the patient in the operating room until the induction of the anesthesia will be controlled by a member of the anesthesia team (regardless of the room process);
  Interventions: Procedure: Control; Procedure: Nursing

INTERVENTIONS:
Procedure: Control — All previously selected patients will be under passive warming by means of blankets
Procedure: Nursing — All previously selected patients will be under active air flow warming device at 43 Celsius

SUMMARY:
Literature establishes that warming with a heated blanket before and during the operation is effective in the prevention of perioperative hypothermia, both in general anesthesia as well as spinal anesthesia. However, the trials have still not presented us with objective protocols to standardize this routine in the surgical centers.

The study aims to assess the adoption and reproduction of the implementation of the warning device by the nursing team immediately after the patient's entrance in the operating room, even before the entrance of the anesthesiologist.

DETAILED DESCRIPTION:
After approval by the Institutional Research Ethics Committee, the patients for elective surgeries to be submitted to general and spinal anesthesia lasting 60 minutes or more held at the central operating center at Santa Casa de Misericórdia in São Paulo will be assessed over a period of 60 days. The patients will receive the necessary explanations on the research and, after obtaining the responsible consent for participating in the trial, they will be included.

Inclusion/exclusion criteria:

Inclusion - adults that will be submitted to general or spinal anesthesia in the central operating center at Santa Casa de Misericórdia in São Paulo.

Exclusion:

* Patient over 18 years old;
* Patients that are feverish/present with infectious symptoms
* Refusal of the use of the device by the patient
* Patient that does not tolerate the use of the blanket in the pre op. The study aims to assess over a period of 60 days the compliance to the protocol and the prewarming time with the use of the heated air flow device from the moment the patients enter the operating room until anesthesia induction. The heating device will be set up connected to the patient and to the motor with the activation of the system at 43°C by the nursing team. The monitoring of the times since the entrance of the patient in the operating room until the induction of the anesthesia will be controlled by a member of the anesthesia team (regardless of the room process).

All the patients scheduled with elective surgery predicted to last over 60 minutes will be selected and there will be an assessment of the number of cases in which the protocol was followed and the time of use of the warming device will be monitored from the installation entrance in the OR and before the anesthesia induction and every 30 minutes beginning of anesthesia, during the surgery until the end of the anesthetic procedure.

The variables to be assessed in the study are:

* Age, gender, weight, height, body mass index (BMI), diseases, physical condition according to the American Anesthesiology Association classification;
* Oral temperature measured at the following points:

  * M-entrance - entering the room and installation of the blanket
  * M-ind - from the moment after the induction of anesthesia;
  * M30, M60, M90, M120 = 30, 60, 90, 120 min after induction till the end of the anesthetic procedure; and the patients scheduled to general anesthesia will be also measured with esophagus thermometer
* The protocol establishes the types of warm blankets available to be used for the different types of surgery;
* Arterial oxygen saturation; heart beat; systolic and diastolic pressure and carbon dioxide expired:

  * At the entrance of the operating room;
  * Immediately after induction;
  * Every 30 minutes after induction until the patient leaves the operating room;
* The type of surgery and anesthesia will be assessed among the pre-warming groups
* Room temperature will be measured (at the entrance of the patient and after induction and at the end of surgery/anesthesia;
* Presence of side effects. The need of blood transfusion will be assessed during surgery. There will be statistical assessment of the results, the significant statistical difference will be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults that will be submitted to general or spinal anesthesia in the surgical center of hospital central at Santa Casa de Misericórdia in São Paulo

Exclusion Criteria:

* Patient under 18 years old;
* Patients that are feverish/present with infectious symptoms
* Refusal of the use of the device by the patient
* Patient that does not tolerate the use of the blanket in the pre op.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Body temperature | 120 minutes
  temperature from entrance in surgical room to ending of anesthesia state

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Caio G De Bernardis, MD, Ph.D, Principal Investigator — Irmandade Santa Casa deMisericórdia de São Paulo
Locations (1):
- Faculdade de Ciencias Medicas da Santa Casa de São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Vaughan MS, Vaughan RW, Cork RC. Postoperative hypothermia in adults: relationship of age, anesthesia, and shivering to rewarming. Anesth Analg. 1981 Oct;60(10):746-51. PMID 7197479
- [Result] Sessler DI. Perioperative thermoregulation and heat balance. Ann N Y Acad Sci. 1997 Mar 15;813:757-77. doi: 10.1111/j.1749-6632.1997.tb51779.x. PMID 9100967
- [Result] Sessler DI, Schroeder M, Merrifield B, Matsukawa T, Cheng C. Optimal duration and temperature of prewarming. Anesthesiology. 1995 Mar;82(3):674-81. doi: 10.1097/00000542-199503000-00009. PMID 7879936
- [Result] Hynson JM, Sessler DI, Glosten B, McGuire J. Thermal balance and tremor patterns during epidural anesthesia. Anesthesiology. 1991 Apr;74(4):680-90. doi: 10.1097/00000542-199104000-00011. PMID 2008950
- [Result] Matsukawa T, Sessler DI, Sessler AM, Schroeder M, Ozaki M, Kurz A, Cheng C. Heat flow and distribution during induction of general anesthesia. Anesthesiology. 1995 Mar;82(3):662-73. doi: 10.1097/00000542-199503000-00008. PMID 7879935
- [Result] Hendolin H, Lansimies E. Skin and central temperatures during continuous epidural analgesia and general anaesthesia in patients subjected to open prostatectomy. Ann Clin Res. 1982 Aug;14(4):181-6. PMID 7168548
- [Result] Insler SR, Sessler DI. Perioperative thermoregulation and temperature monitoring. Anesthesiol Clin. 2006 Dec;24(4):823-37. doi: 10.1016/j.atc.2006.09.001. PMID 17342966
- [Result] Kurz A, Sessler DI, Christensen R, Dechert M. Heat balance and distribution during the core-temperature plateau in anesthetized humans. Anesthesiology. 1995 Sep;83(3):491-9. doi: 10.1097/00000542-199509000-00007. PMID 7661349
- [Result] Hynson JM, Sessler DI, Moayeri A, McGuire J, Schroeder M. The effects of preinduction warming on temperature and blood pressure during propofol/nitrous oxide anesthesia. Anesthesiology. 1993 Aug;79(2):219-28, discussion 21A-22A. doi: 10.1097/00000542-199308000-00005. PMID 8342834
- [Result] Sessler DI, Moayeri A. Skin-surface warming: heat flux and central temperature. Anesthesiology. 1990 Aug;73(2):218-24. PMID 2382847
- [Result] Neubauer RA, James P. Cerebral oxygenation and the recoverable brain. Neurol Res. 1998;20 Suppl 1:S33-6. doi: 10.1080/01616412.1998.11740606. PMID 9584921
- [Result] Vanni SM, Braz JR, Modolo NS, Amorim RB, Rodrigues GR Jr. Preoperative combined with intraoperative skin-surface warming avoids hypothermia caused by general anesthesia and surgery. J Clin Anesth. 2003 Mar;15(2):119-25. doi: 10.1016/s0952-8180(02)00512-3. PMID 12719051
- [Result] Kurz A, Kurz M, Poeschl G, Faryniak B, Redl G, Hackl W. Forced-air warming maintains intraoperative normothermia better than circulating-water mattresses. Anesth Analg. 1993 Jul;77(1):89-95. doi: 10.1213/00000539-199307000-00018. PMID 8317754
- [Result] Matsuzaki Y, Matsukawa T, Ohki K, Yamamoto Y, Nakamura M, Oshibuchi T. Warming by resistive heating maintains perioperative normothermia as well as forced air heating. Br J Anaesth. 2003 May;90(5):689-91. doi: 10.1093/bja/aeg106. PMID 12697600
- [Result] Torrie JJ, Yip P, Robinson E. Comparison of forced-air warming and radiant heating during transurethral prostatic resection under spinal anaesthesia. Anaesth Intensive Care. 2005 Dec;33(6):733-8. doi: 10.1177/0310057X0503300605. PMID 16398377
- [Result] Hynson JM, Sessler DI. Intraoperative warming therapies: a comparison of three devices. J Clin Anesth. 1992 May-Jun;4(3):194-9. doi: 10.1016/0952-8180(92)90064-8. PMID 1610573
- [Result] Horn EP, Bein B, Bohm R, Steinfath M, Sahili N, Hocker J. The effect of short time periods of pre-operative warming in the prevention of peri-operative hypothermia. Anaesthesia. 2012 Jun;67(6):612-7. doi: 10.1111/j.1365-2044.2012.07073.x. Epub 2012 Feb 29. PMID 22376088